CLINICAL TRIAL: NCT00795613
Title: Multicenter Clinical Study With Early Treatment Intensification In Patients With High- Risk Hodgkin Lymphoma, Identified As FDG-PET Scan Positive After 2 Conventional ABVD Courses
Brief Title: Positron Emission Tomography (PET)-Adapted Chemotherapy In Advanced Hodgkin Lymphoma (HL)
Acronym: HD0607
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ospedale Santa Croce-Carle Cuneo (Other)
Collaborators: GITIL (GRUPPO ITALIANO TERAPIE INNOVATIVE NEI LINFOMI) (Unknown); Consorzio Mario Negri Sud (Other)
Responsible Party: Principal Investigator, DR. ANDREA GALLAMINI, HEAD OF HAEMATOLOGY DEPT. A.S.O. S. CROCE AND CARLE, Ospedale Santa Croce-Carle Cuneo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GITIL - HD0607
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: HODGKIN LYMPHOMA
Keywords: PET
MeSH Terms: conditions — Hodgkin Disease | interventions — Etoposide; Cyclophosphamide; Procarbazine; deltacortene; Rituximab; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PET pos (Experimental): Patients With Interim Pet Positive Proceed To Escalated Beacopp Regimen
  Interventions: Drug: ESCALATED BEACOPP
- PET negative (Other): Patients With Interim-Pet Negative Continue The Conventional ABVD Regimen
  Interventions: Drug: CONVENTIONAL ABVD

INTERVENTIONS:
Drug: ESCALATED BEACOPP — Esc.BEACOPP Bleomicine10 mg/m2/ev/die 8° VP-16 200 mg/m2/ev/die1°- 3° Doxorubicine35 mg/m2/ev/die 1° Cyclophosphamide1250 mg/m2/ev/die 1° Vincristine1,4 mg/m2(max dose 2 mg)/ev/die 8° Procarbazine100 mg/m2/b.m./die 1°- 7° Prednison40 mg/m2/b.m./die 1°-14° G-CSF300mcg/die s/c from day 8 until PMN>1000/ul Recycle every 21 days Esc.R-BEACOPP as above plus Rituximab 375 mg/m2/ev/ die 1° Recycle every 21 days Baseline BEACOPP Bleomicine10 mg/m2/ev/die 8° VP-16 100 mg/m2/ev/die 1°-3° Doxorubicine25 mg/m2/ev/die 1° Cyclophosphamide650 mg/m2/ev/die 1° Vincrinstine1,4 mg/m2(max dose 2 mg)/ev/die 8° Procarbazine100 mg/m2/os/die 1°-7° Prednison40 mg/m2/os/die 1°-14° Recycle every 21 days Baseline R-BEACOPP as above plus Rituximab375 mg/m2/ev/ die 1° Recycle every 21 days
  Other Names: BLEOMICINE TEVA; VEPESID; DOXORUBICINE TEVA; ENDOXAN; VINCRISTINE TEVA; NATULAN; DELTACORTENE; MABTHERA
  Arms: PET pos
Drug: CONVENTIONAL ABVD — ABVD(cycle repeats every 28 days) Doxorubicine25 mg/m2 iv days 1,15 Bleomicine10,000 units/m2 iv days 1,15 Vinblastine6 mg/m2 iv days 1,15 Dacarbazine375mg/m2 iv days 1,15 This will be given at full dose and on schedule,regardless of blood count.
  Other Names: BLEOMICINE TEVA; DOXORUBICINE TEVA; VELBE; NATULAN
  Arms: PET negative

SUMMARY:
The purpose of this multicenter clinical trial is to assess the clinical impact of dose intensification performed very early during treatment in a subset of poor prognosis, advanced-stage Hodgkin Lymphoma patients, defined as PET-positive after two courses of conventional adriamycin (doxorubicin), bleomycin, vinblastine and dacarbazine (ABVD) chemotherapy.

DETAILED DESCRIPTION:
Version number 1.0 Date 07.05.0808

Study Title

A phase-II clinical trial for assessing the clinical impact of a global strategy utilizing early FDG-PET imaging for a risk-adapted therapy in untreated, advanced Hodgkin Lymphoma (aHL).

Short study title PET-adapted chemotherapy in advanced HL

Start and end dates of study Start date: July 2008

Patients will be recruited during four calendar years and will be followed at least for three years.

Registration of the patients All patients with newly diagnosed Hodgkin's Lymphoma, presenting with advanced disease (stage II B-IV B) should be registered at the WEB site of the study whatever treatment is planned.

Primary outcome measure 3-year progression free survival (PFS).

Secondary endpoint 3-year event free survival (EFS) of all the registered patients whatever the treatment assigned. Events are deaths from any cause, disease progression, secondary cancer, late serious treatment-related events.

- Feasibility of the program for the entire population of advanced-stage HL patients admitted to GITIL institutions

Clinical Phase Phase II

Study design A multicentre clinical trial for assessing the clinical impact of a global strategy utilizing early FDG-PET imaging after 2 cycles of ABVD for a risk-adapted, single patient tailored therapy for all the newly diagnosed, aHL patients admitted to GITIL haematological centers .

Statistical aspects 450 patients could be recruited in GITIL centres in 4 years. Thirty-five percent of these could be expected to have a PET-2 positive after 2 ABVD courses (135 patients). Roughly half of these latter could likely be salvaged by BEACOPPescal. or R-BEACOPPescal. therapy. Since the 3-y PFS of aHL patients treated with the ABVD is 70% we could expect to cure, with this approach, about 85% of these patients. In order to demonstrate a benefit of this strategy over conventional ABVD treatment, with the Simon optimal two-stage design and an alpha error of 0.05 and a power of 90%, a minimum of 150 patients needs to be enrolled. In order to establish an advantage of R-BEACOPP esc. over BEACOPPescal. Approximately 135 patients are needed in the arm of PET-positive patients.

Analysis will be intention-to-treat. Standard time-to-event statistics tests will be carried out, including Kaplan-Meier survival curves, log rank test, and Cox proportional hazards models. Chi square test and analysis of variance will be adopted for univariate analysis with mathematical transformation to approach normality as appropriate. The formal level of significance for P-values is set at 0.05 (two-tailed).

Interim analysis and safety aspects A first interim analysis is planned one year after study onset in order to check the morbidity and mortality of the program. Because of the rarity of the disease, no formal statistical boundaries are established as stopping rules. The results of the interim analysis will be evaluated by the Data Safety and Monitoring Board (DSMB). The Chairman of the DSMB will advise the Steering Committee (ST) as to the any action to be taken for safety reasons (i.e., premature study closure and protocol modification). The DSMB will also establish and communicate to the ST and the CRO its own rules and requirements to optimize the quantity and quality of information to be periodically received to monitor adequately all safety aspects.

Initial treatment for 2 cycles ABVD (cycle repeats every 28 days) This will be given at full dose and on schedule, regardless of blood count. Growth factors may be used at the discretion of investigators but are not routinely advised.

PET Reviewing Committee A central panel for PET reviewing (PET-RC) will be established. The members will be seven nuclear medicine experts. The operational aspects of the validation of PET diagnoses will be managed by the National Institute of Nuclear Physics in Turin using an already existing and functioning web-site. Upon receipt of PET-2 records, along with PET baseline studies via web, the PET-RC members are bound to send the reviewed studies to the Central Data Center (CDC) within 5 days from the data of receipt of the studies from the local PET enter. The image exchange will be performed by uploading the records of PET-2 (PET after 2 cycles of ABVD) and PET-0 (baseline PET) in the .dycom format in the web site dedicated.Only the positive and "minimally positive" PET scan will be reviewed. The final judgment of a reviewed defined as "positive" or "negative" study will be supplied from the CDC to the local GITIL center on the basis of the first three reviewed studies arrived to CDC

After 2 cycles, PET negative patients (Arm B) continue with ABVD (for 4 cycles) ABVD as above, every 28 days for 4 further cycles Patients in Arm B with a positive PET at the end of ABVD treatment. Patients with a positive PET at the end of ABVD chemotherapy should undergo, whenever is possible, a confirmatory biopsy; in patients with a proven resistant disease DHAP (x1 or x2) should be given in order to collect a sufficient number of CD 34+ cells; later they proceed to a classical high-dose sequential chemotherapy (HDS) with: cyclophosphamide 4 gr./m2 , ARA-c 4 gr./m2/day for 4 days, VP 16 2 gr./m2, followed by autologous stem cell transplantation (ASCT) with BEAM conditioning regimen

Consolidation Radiotherapy (Arm B) Patients treated with traditional ABVD x 6 cycles (PET-negative arm) will be re-evaluated at the end of chemotherapy with PET. Patients with a negative final PET scan will be randomized to undergo consolidation radiotherapy or not on the initial bulky lesion(s) or on the residual disease. Radiotherapy will be given with an "involved field technique, at the dose of 30 Gy. No radiotherapy is planned in patients with residual mass that was not an initial bulky lesion.

After 2 cycles, PET positive patients (Arm A) will be randomized to 4 escalated BEACOPP or 4 escalated R-BEACOPP administration for 4 cycles. Peripheral Blood Stem Cell (PBSC) will be collected after the first BEACOPP (or R-BEACOPP) course

After 4 cycles of escalated BEACOPP or escalated R-BEACOPP patients with PET negative will continue with baseline BEACOPP or baseline R-BEACOPP (for further 4 cycles )

After 4 cycles of escalated BEACOPP or escalated R-BEACOPP patients with positive PET will undergo salvage treatment with DHAP (x 1 or x 2) followed by double autologous stem cell transplantation (ASCT) or, in presence of a suitable HLA-matched stem cell donor, with a single ASCT (BEAM) followed by RIC allogeneic bone marrow transplantation .

Allogeneic Reduced-Intensity transplant:

Thiotepa 5 mg/Kg every 12 hours for 2 doses (day -5); cyclophosphamide 30 mg/kg (days -4 and -3); fludarabine 30 mg/ms (days -4 and -3); allogeneic stem cell transplantation with 4 - 8 X 106 CD34+ cells/kg from related donors (day 0).

GVHD prophylaxis:

Cyclosporin A (CSA), adjusted to 200-300 ng/ml blood levels, and short course methotrexate (10 mg/ms day +1, 8 mg/ms day + 3 and +6). CSA is administered at full dose through day +100 and, if GVHD does not occur, the dose is tapered by 10% every week thereafter

Treatment duration Approx 10-11 months for PET-2+ patients and 6 months for PET-2 negative patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced classical Hodgkin Lymphoma according to the World Health Organization classification
* Aged 18-60
* Not previously treated
* Stages IIB to IV B
* All IPS prognostic groups
* Patients who have signed an informed consent form

Exclusion Criteria:

* Patients aged more than 60.
* Concomitant or previously treated neoplastic disorder less than 5 year before the diagnosis of Hodgkin's lymphoma.
* Psychiatric disorders
* Uncontrolled infectious disease
* Impaired cardiac (EF < 50%) , renal (creatinine clearance < 60 ml/m)
* HIV, HBV DNA, HCV RNA positive markers
* Pregnancy and lactation
* Patients with uncompensated diabetes mellitus and fasting glucose levels over 200 mg/dl

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2008-06; Primary Completion 2014-11 (Actual); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 3 year

SECONDARY OUTCOMES:
event-free survival (EFS) | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: ANDREA GALLAMINI, MD, Study Chair — A.S.O. S.CROCE E CARLE-HEMATOLOGY DEPT. - VIA M. COPPINO 26-12100 CUNEO ITALY
Locations (24):
- The Chaim Sheba Medical Center, Tel Litwinsky, Israel
- Italy (23):
  - Ospedale S. Gerardo, Monza, Milano
  - A.O. Universitaria S. Luigi Gonzaga, Orbassano, Torino
  - A.O. Universitaria Ospedali Riuniti Osp. Umberto I, Ancona
  - Ospedali Riuniti, Bergamo
  - Ospedale Generale Regionale Bolzano, Bolzano
  - Ospedale Roberto Binaghi, Cagliari
  - A.O. Universitaria Osp. Vittorio Emanuele E Ferrarotto, Catania
  - Azienda Ospedaliera S. Croce E Carle, Cuneo
  - Azienda Ospedaliera Universitaria S. Martino, Genova
  - Ospedale S. Raffaele Turro, Milan
  - Irccs - Istituto Nazionale Dei Tumori (Int), Milan
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan
  - A.O. Universitaria Federico Ii, Napoli
  - Azienda Ospedaliera, Padua
  - Azienda Ospedaliera V. Cervello, Palermo
  - Ospedale Silvestrini-S.Andrea Delle Fratte, Perugia
  - Ospedale S. Carlo, Potenza
  - A.O. Universitaria Policlinico Tor Vergata, Roma
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - Ospedale Mauriziano Umberto I, Torino
  - A.O. Universitaria S. Giovanni Battista-Molinette, Torino
  - Ospedale Policlinico G.B. Rossi, Verona
  - Ospedale Di Vicenza, Vicenza

REFERENCES:
- [Background] Gallamini A, Hutchings M, Rigacci L, Specht L, Merli F, Hansen M, Patti C, Loft A, Di Raimondo F, D'Amore F, Biggi A, Vitolo U, Stelitano C, Sancetta R, Trentin L, Luminari S, Iannitto E, Viviani S, Pierri I, Levis A. Early interim 2-[18F]fluoro-2-deoxy-D-glucose positron emission tomography is prognostically superior to international prognostic score in advanced-stage Hodgkin's lymphoma: a report from a joint Italian-Danish study. J Clin Oncol. 2007 Aug 20;25(24):3746-52. doi: 10.1200/JCO.2007.11.6525. Epub 2007 Jul 23. PMID 17646666
- [Background] Gallamini A, Rigacci L, Merli F, Nassi L, Bosi A, Capodanno I, Luminari S, Vitolo U, Sancetta R, Iannitto E, Trentin L, Stelitano C, Tavera S, Biggi A, Castagnoli A, Versari A, Gregianin M, Pelosi E, Torchio P, Levis A. The predictive value of positron emission tomography scanning performed after two courses of standard therapy on treatment outcome in advanced stage Hodgkin's disease. Haematologica. 2006 Apr;91(4):475-81. PMID 16585014
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] Gallamini A, Rossi A, Patti C, Picardi M, Romano A, Cantonetti M, Oppi S, Viviani S, Bolis S, Trentin L, Gini G, Battistini R, Chauvie S, Sorasio R, Pavoni C, Zanotti R, Cimminiello M, Schiavotto C, Viero P, Mule A, Fallanca F, Ficola U, Tarella C, Guerra L, Rambaldi A. Consolidation Radiotherapy Could Be Safely Omitted in Advanced Hodgkin Lymphoma With Large Nodal Mass in Complete Metabolic Response After ABVD: Final Analysis of the Randomized GITIL/FIL HD0607 Trial. J Clin Oncol. 2020 Nov 20;38(33):3905-3913. doi: 10.1200/JCO.20.00935. Epub 2020 Sep 18. PMID 32946355
- [Derived] Gallamini A, Tarella C, Viviani S, Rossi A, Patti C, Mule A, Picardi M, Romano A, Cantonetti M, La Nasa G, Trentin L, Bolis S, Rapezzi D, Battistini R, Gottardi D, Gavarotti P, Corradini P, Cimminiello M, Schiavotto C, Parvis G, Zanotti R, Gini G, Ferreri AJM, Viero P, Miglino M, Billio A, Avigdor A, Biggi A, Fallanca F, Ficola U, Gregianin M, Chiaravalloti A, Prosperini G, Bergesio F, Chauvie S, Pavoni C, Gianni AM, Rambaldi A. Early Chemotherapy Intensification With Escalated BEACOPP in Patients With Advanced-Stage Hodgkin Lymphoma With a Positive Interim Positron Emission Tomography/Computed Tomography Scan After Two ABVD Cycles: Long-Term Results of the GITIL/FIL HD 0607 Trial. J Clin Oncol. 2018 Feb 10;36(5):454-462. doi: 10.1200/JCO.2017.75.2543. Epub 2018 Jan 23. PMID 29360414